CLINICAL TRIAL: NCT07342634
Title: Effect of Blood Flow Restriction on Recovery After Maximal Resistance Exercise: a Controlled Clinical Trial
Brief Title: Effect of Blood Flow Restriction on Recovery After Maximal Resistance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Principal Investigator, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 91529125.6.0000.5402
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Recovery; Recovery Time
Keywords: Resistance training; physiological stress; post-exercise recovery; blood flow restriction therapy; functional physical performance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blood flow restriction with 80% occlusion (Experimental): Will perform an BFR intervention using 80% of the total occlusion pressure (TOP) continuously for 20 minutes.
  Interventions: Device: BFR-80%
- Blood flow restriction with 60% occlusion (Experimental): Will perform an BFR intervention using 60% of the total occlusion pressure (TOP) continuously for 20 minutes.
  Interventions: Device: BFR-60%
- Blood flow restriction with 10 mmHg of occlusion pressure (Placebo Comparator): The intervention will be performed with BFR using 10 mmHg of occlusion pressure continuously for 20 minutes.
  Interventions: Other: BFR-10mmHg
- Control (No Intervention): It will remain at rest for 20 minutes without using BFR.

INTERVENTIONS:
Device: BFR-80% — Will perform the intervention with BFR using 80% of the total occlusion pressure (TOP) continuously for 20 minutes.
  Arms: Blood flow restriction with 80% occlusion
Device: BFR-60% — Will perform the intervention with BFR using 60% of the total occlusion pressure (TOP) continuously for 20 minutes.
  Arms: Blood flow restriction with 60% occlusion
Other: BFR-10mmHg — Will perform the intervention with BFR using 10 mmHg of occlusion pressure continuously for 20 minutes.
  Arms: Blood flow restriction with 10 mmHg of occlusion pressure

SUMMARY:
Resistance training has been widely performed due to its health benefits. However, performing this training at high intensity causes significant muscle stress, leading to fatigue and compromising performance. It is essential to implement effective recovery strategies to optimize physiological adaptations. Among the accessible techniques, blood flow restriction (BFR) has shown promise for its potential to accelerate muscle recovery.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted with 40 men and 40 women allocated to one of four groups: i) BFR using 80% of total occlusion pressure (TOP) [BFR-80%]; ii) BFR using 60% of total occlusion pressure (TOP) [BFR-60%]; iii) BFR using 10 mmHg (BFR-10 mmHg); and iv) control (CON). All groups will undergo initial assessments, followed by the muscle stress protocol, and all outcomes will be collected again. Subsequently, the intervention to which they were previously randomized will be performed, and finally, subsequent assessments will be conducted immediately, 24, 48, and 72 hours after exercise. The outcomes assessed will be, in order: pain using the Numerical Rating Scale (NRS), perception of recovery and discomfort using the Likert scale, and perception of effort using the Borg scale (CR-10), cellular integrity vectors using bioelectrical impedance analysis (BIA), pain threshold using a pressure algometer, muscle tone, stiffness, and elasticity using myotonometry, quadriceps muscle strength test using a digital dynamometer, muscle power test using the Squat Jump test, and a single-leg jump functional test.

Participants will be duly informed about the procedures and objectives of this study, and after agreeing, will sign a free and informed consent form, thus becoming effectively part of it. In the consent form, participants will be asked if they agree to the use of their data should they choose to withdraw from the study. Participants will also be asked for permission for the research team to share relevant data with people from the universities participating in the research or regulatory authorities, when relevant, while preserving the participant's identity. The study will be submitted for review and approval to the Research Ethics Committee of FCT/UNESP, Presidente Prudente, SP, Brazil and will be registered on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Individuals exhibiting one or more of the following characteristics will not be included:
* (1) diabetes and hypertension;
* (2) inflammatory rheumatological, psychiatric, cardiovascular and/or respiratory disease;
* (3) pre-existing injury restricting their ability to perform vigorous physical activities;
* (4) having one or more predisposing risk factors for thromboembolism.

Exclusion Criteria:

* Participants will be excluded from the study if they:
* (1) have a health problem that does not allow them to continue;
* (2) wish to leave the study;
* (3) use medications, electrotherapy, or other therapeutic methods during the study period that could interfere with any results;
* (4) not sign the consent form.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lower limb muscle power | Change from baseline at 72 hours after exercise
  Muscle power will be assessed through the Squat Jump test using a contact platform (Multisprint). Participants will begin in a 90° knee flexion position (verified with a goniometer), with hands on hips, and will perform a vertical jump without countermovement. Variables to be analyzed will include jump height, modified reactive strength index, jump power, and take-off moment.
Lower limb muscle function | Change from baseline at 72 hours after exercise
  Muscle function will be assessed through the single leg hop functional test sing a measuring tape in centimeters. The participant will be positioned standing on a flat surface, barefoot, and with their hands on their waist. They will be asked to perform a horizontal jump with the greatest possible reach using only one lower limb (test performed unilaterally). The contralateral limb will remain flexed without touching the ground during the execution. After the jump, the participant must maintain balance for at least two seconds without losing stability or moving the landing foot. The jump distance will be measured in centimeters from the toe of the supporting foot (before the jump) to the heel at the moment of landing, using a measuring tape.
Isometric strenght of quadriceps and hamstring muscle | Change from baseline at 72 hours after exercise
  The isometric peak torque of the quadriceps and hamstring will be measured using a digital handheld dynamometer (DD-300, Instrutherm). For the quadriceps strength assessment, the participant will be seated in a chair with their knee bent at 90° and instructed to push maximally against the dynamometer. To measure hamstring strength, the participant will be positioned in a prone position with their knee flexed at 90º and will be instructed to push maximally against the dynamometer. Three attempts will be performed with a 1-minute rest interval. The highest value will be used for analysis.
Muscle soreness and pain threshold | Change from baseline at 72 hours after exercise
  Muscle soreness will be assessed using a Numeric Pain Rating Scale (0-10). Pain threshold will be measured with a pressure algometer (FPX 50/220; Wagner) at four sites: biceps femoris and rectus femoris. Measurements will be recorded in kgf and will not exceed 2.55 kgf.
Perceived exertion, recovery, and discomfort | Change from baseline at 72 hours after exercise
  Perceived exertion, recovery, and discomfort will be measured using the Borg CR-10 scale (0-10). Participants will rate: (1) exertion as whole-body effort, (2) discomfort as muscular sensations in the lower limbs, and (3) recovery as general physical and psychological recovery. Values will be individually recorded at each time point.
Myotonometry | Change from baseline at 72 hours after exercise
  Muscle tone, stiffness, and elasticity will be measured using the MyotonPRO device. The probe will be positioned perpendicularly over the following sites: biceps femoris and rectus femoris. The device will apply a 0.18 N pre-load and a 0.40 N impulse to induce tissue oscillation for measurement.
Bioelectrical impedance analysis | Change from baseline at 72 hours after exercise
  Bioimpedance will be measured using a tetrapolar device (BIA Analyzer, 50 kHz, 800 µA). Electrodes will be positioned on the biceps femoris and rectus femoris. Analyzed variables will include resistance (R), reactance (Xc), phase angle (PhA), and tolerance ellipse, via Bioscan software.

OTHER OUTCOMES:
Occlusion pressures (AOP) | Baseline
  To determine the AOP, the Doppler equipment transducer will be used, which will be positioned over the posterior tibial artery to capture the auscultatory pulse. A blood pressure cuff will be fixed to the participant's thigh close to the region of the inguinal fold of the dominant limb, and then with the inflatable region of the cuff on the medial portion of the thigh covering the femoral artery, it will be progressively inflated, waiting 15 seconds every 30 mmHg until the point at which the auscultatory pulse of the tibial artery is interrupted.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No